CLINICAL TRIAL: NCT00864097
Title: A PHASE 3, RANDOMIZED, DOUBLE BLIND, CONTROLLED, MULTI CENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB ADDED ON TO DICLOFENAC SR IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: Analgesic Efficacy And Safety of Tanezumab Added On To Diclofenac SR In Patients With Osteoarthritis Of The Knee Or Hip
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091017; 2009-009318-41 (EudraCT Number); P3 6 MO OA HIP/KNEE DICLOFENAC (Other: Alias Study Number)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis
Keywords: Arthritis monoclonal antibody nerve growth factor (NGF) anti-NGF tanezumab PF-04383119 RN-624 OA
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tanezumab 10 mg + diclofenac (Experimental): IV tanezumab 10 mg every 8 weeks (through Week 16) and oral diclofenac SR 75 mg BID (through Week 32)
  Interventions: Biological: tanezumab; Drug: diclofenac
- Tanezumab 5 mg + diclofenac (Experimental): IV tanezumab 5 mg every 8 weeks (through Week 16) and oral diclofenac SR 75 mg BID (through Week 32)
  Interventions: Biological: tanezumab; Drug: diclofenac
- Tanezumab 2.5 mg + diclofenac (Experimental): IV tanezumab 2.5 mg every 8 weeks (through Week 16) and oral diclofenac SR 75 mg BID (through Week 32)
  Interventions: Biological: tanezumab; Drug: diclofenac
- IV placebo + diclofenac (Placebo Comparator): IV placebo to match tanezumab every 8 weeks (through Week 16) and oral diclofenac SR 75 mg BID (through Week 32)
  Interventions: Drug: diclofenac; Other: IV placebo

INTERVENTIONS:
Biological: tanezumab — IV tanezumab 10 mg every 8 weeks (through Week 16)
  Arms: Tanezumab 10 mg + diclofenac
Drug: diclofenac — Oral diclofenac SR 75 mg BID for 32 weeks
  Arms: Tanezumab 10 mg + diclofenac
Biological: tanezumab — IV tanezumab 5 mg every 8 weeks (through Week 16)
  Arms: Tanezumab 5 mg + diclofenac
Drug: diclofenac — Oral diclofenac SR 75 mg BID for 32 weeks
  Arms: Tanezumab 5 mg + diclofenac
Biological: tanezumab — IV tanezumab 2.5 mg every 8 weeks (through Week 16)
  Arms: Tanezumab 2.5 mg + diclofenac
Drug: diclofenac — Oral diclofenac SR 75 mg BID for 32 weeks
  Arms: Tanezumab 2.5 mg + diclofenac
Drug: diclofenac — Oral diclofenac SR 75 mg BID for 32 weeks
  Arms: IV placebo + diclofenac
Other: IV placebo — IV placebo to match tanezumab every 8 weeks (through Week 16)
  Arms: IV placebo + diclofenac

SUMMARY:
The purpose of this study is to investigate the analgesic efficacy and safety of tanezumab added on to diclofenac SR in patients with osteoarthritis of the knee or hip currently experiencing partial benefit from, and are tolerating, diclofenac 150 mg/day therapy.

DETAILED DESCRIPTION:
This study was terminated on 16 Nov 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip according to ACR criteria with Kellgren-Lawrence X-ray grade equal to, or greater than, 2.
* Patients must be experiencing some benefit from their current stable dose regimen of oral diclofenac 150 mg/day and be tolerating their diclofenac regimen.
* Pain and function levels as required by the protocol at Screening and Baseline.
* Willing to discontinue all non-study pain medications throughout the study except as permitted per protocol.
* Willing and able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Pregnant women.
* BMI greater than 39.
* History of other disease that may involve index knee or hip including inflammatory joint diseases, chrystalline disease (gout or pseudogout), endocrinopathies, metabolic joint diseases, lupus erythematosus, rheumatoid arthritis (RA), joint infections, neuropathic disorders, avascular necrosis, Paget's disease or tumors.
* Fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy or other moderate to severe pain that may confound assessments or self-evaluation of the pain associated with OA.
* Signs and symptoms of clinically significant cardiac disease within 6 months prior to screening.
* Diagnosis or TIA within 6 months prior to screening or diagnosis of stroke with residual deficits that would preclude completion of required study activities.
* History, diagnosis , signs or symptoms of clinically significant neurological and/or psychiatric disease/disorder.
* At Screening: uncontrolled hypertension, hemoglobin A1c greater than or equal to 10%, ALT or AST greater than or equal to 3X upper limit of normal, creatinine exceeding 150 micro-mol/L in men or 133 micro-mol/L in women.
* Patients on warfarin or other coumadin anticoagulant therapy and/or lithium therapy within 30 days prior to Screening.
* Known hypersensitivity to NSAIDs (eg, diclofenac), cyclooxygenase inhibitors or paracetamol (acetaminophen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2009-08-11 (Actual); Primary Completion 2010-11-16 (Actual); Study Completion 2010-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- Austria (5):
  - LKH-Medizinische Universitatsklinik Graz, Graz
  - Nuhr Zentrum, Senftenberg
  - ClinPharm International GmbH, Vienna
  - Medizinische Universitaet Wien/AKH, Vienna
  - Rheuma Zentrum Favoriten, Vienna
- France (2):
  - CHU de Nantes, Nantes
  - Hopital Lariboisiere, Paris
- Germany (21):
  - Charité-Universitaetsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Apotheke, Berlin
  - Herz Apotheke, Bochum
  - Synexus ClinPharm GmbH, Bochum
  - Viereck-Apotheke, Buch
  - Synexus ClinParm GmbH, Dresden
  - Apotheke im Arztehaus Mickten, Dresden
  - Schiller Apotheke & Stadt Apotheke, Göppingen
  - Schmerz- und Palliativzentrum Goeppingen, Göppingen
  - Falken Apotheke Hoheluft, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover - Mitte GmbH, Hanover
  - Loewen-Apotheke, Hanover
  - Synexus ClinPharm GmbH, Leipzig
  - Arkana Apotheke OHG, Leipzig
  - Synexus ClinPharm GmbH, Magdeburg
  - Apotheke im MSZ, Magdeburg
  - Apotheke des Ernst von Bergmann Klinikums, Potsdam
  - Synexus ClinParm GmbH, Potsdam
  - Kirchsteig Apotheke, Potsdam
- Poland (5):
  - "Centrum Medyczne MEDENS S.C. Niepubliczny Zaklad, Chełm Śląski
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Centrum Medyczne OSTEOMED Sp. z o. o., Warsaw
  - Synexus SCM Sp. z o.o., Wroclaw
  - Niepubliczny Zaklad Opieki Zdrowotnej "POLIMEDICA", Zgierz
- Romania (8):
  - Municipal Hospital No. 1 "Schuller", Ploieşti, Prahova
  - Clinical Emergency Military Hospital "Dr. Carol Davila", Bucharest
  - Duo Medical srl, Bucharest
  - Medical Center "SANA", Bucharest
  - Clinical Hospital "Sf. Maria", Bucharest
  - Center of Rheumatology "Dr Ion Stoia", Bucharest
  - Clinical Emergency County Hospital Constanta, Constanța
  - County Emergency Clinic Hospital "Sf. Apostol Andrei", Galati
- Russia (8):
  - Center polyclinic of Federal State Institution, Arkhangelsk
  - State Healthcare Institution of Moscow city "City Clinical Hospital #15 n.a. O. M. Filatov", Moscow
  - Chair of Hospital Therapy of Ryazan State Medical University, Ryazan
  - St. Petersburg State Healthcare Institution "City Hospital #25 City Rheumatology Center", Saint Petersburg
  - State Educational Institution of Additional Professional Education, Saint Petersburg
  - Institution of Russian Academy of Sciences "St. Petersburg Clinical Hospital of RAS", Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Outpatient Clinical #51", Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Pokrovskaya Hospital", Saint Petersburg
- Spain (7):
  - Hospital Nuestra Señora de la Esperanza, Santiago de Compostela, A Coruna
  - Centro Salud Petrer 1, Petrel, Alicante
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Comarcal de Elda, Elda Alicante
  - Hospital Universitario Getafe, Getafe-Madrid
  - Hospital G. U. Gregorio Maranon, Madrid
  - Hospital Clinico Universitario Santiago, Santiago de Compostela
- Sweden (3):
  - Me3plus AB, Gothenburg
  - Center for Lakemedelsstudier, Malmo
  - Medicinskt Centrum, Norrköping
- Ukraine (14):
  - Chernivtsi Regional Clinical Hospital,Department of Rheumatology, Chernivtsi
  - Road Clinical Hospital at Dnipropetrovsk station, Department of Rheumatology, Dnipropetrovsk
  - Institute of Urgent and Recovery Surgery named after V.K. Gusaka AMS Ukraine, Donetsk
  - Central City Clinical Hospital#1, Department of Therapy,, Donetsk
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - City Clinical Hospital #8, Department of reumatology,, Kharkiv
  - State Institution "Institute of Gerontology AMS of Ukraine", Kiev
  - Oleksandrivska Clinical Hospital in Kyiv-Department of Rheumatology # 1, Kyiv
  - Kyiv Central Basin Clinical Hospital, Department of cardiology,, Kyiv
  - 4th City Communal Clinical Hospital, Department of Rheumatology,, Lviv
  - City communal clinical hospital #5, Dept. of Therapy, Danylo Galytskiy Lviv National Med. University, Lviv
  - Communal Institution Ternopil regional council, "Ternopil Regional Clinical Hospital", Ternopil
  - Vinnytsya regional clinical hospital named after M.I. Pyrogova, Vinnytsia
  - Communal institution "City Hospital #7", Department of Therapy,, Zaporizhzhia
- United Kingdom (3):
  - Barnsley Hospital NHS Trust, Barnsley, South Yorkshire
  - Department of Rheumatology, Dudley, West Midlands
  - Wrightington Hospital, Wigan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- [Derived] Balanescu AR, Feist E, Wolfram G, Davignon I, Smith MD, Brown MT, West CR. Efficacy and safety of tanezumab added on to diclofenac sustained release in patients with knee or hip osteoarthritis: a double-blind, placebo-controlled, parallel-group, multicentre phase III randomised clinical trial. Ann Rheum Dis. 2014 Sep;73(9):1665-72. doi: 10.1136/annrheumdis-2012-203164. Epub 2013 Jul 12. PMID 23852695
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091017&StudyName=Analgesic%20Efficacy%20And%20Safety%20of%20Tanezumab%20Added%20On%20To%20Diclofenac%20SR%20In%20Patients%20With%20Osteoarthritis%20Of%20The%20Knee%20Or%20Hip

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with osteoarthritis of knee or hip who were receiving and tolerating stable dose of diclofenac 150 milligram (mg) per day but required additional pain relief were recruited in this study.
Pre-assignment Details: After screening, participants received study supplied diclofenac slow release (SR) 75 mg tablet twice daily for a minimum of 14 days prior to randomization.
Groups:
- Placebo + Diclofenac: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion at Baseline, Week 8 and Week 16 along with diclofenac 75 milligram (mg) slow release tablet orally twice daily up to Week 32.
- Tanezumab 2.5 mg + Diclofenac: Tanezumab (RN624 or PF-04383119) 2.5 mg intravenous infusion at Baseline, Week 8 and Week 16 along with diclofenac 75 mg slow release tablet orally twice daily up to Week 32.
- Tanezumab 5 mg + Diclofenac: Tanezumab (RN624 or PF-04383119) 5 mg intravenous infusion at Baseline, Week 8 and Week 16 along with diclofenac 75 mg slow release tablet orally twice daily up to Week 32.
- Tanezumab 10 mg + Diclofenac: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion at Baseline, Week 8 and Week 16 along with diclofenac 75 mg slow release tablet orally twice daily up to Week 32.
Period: Overall Study
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Started | 154 | 157 | 151 | 145
Treated | 152 | 157 | 150 | 145
Completed | 15 | 20 | 19 | 20
Not Completed | 139 | 137 | 132 | 125
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Adverse Event | 6 | 8 | 11 | 9
Not completed — Lack of Efficacy | 9 | 3 | 7 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 11 | 11 | 12
Not completed — Protocol Violation | 2 | 1 | 0 | 1
Not completed — Terminated by sponsor | 105 | 112 | 102 | 99
Not completed — Randomized but not treated | 2 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac | Total
Number analyzed (Participants) | 152 | 157 | 150 | 145 | 604
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 4 | 6 | 4 | 1 | 15
  45 to 64 years | 84 | 86 | 88 | 78 | 336
  Greater than or equal to (>=) 65 years | 64 | 65 | 58 | 66 | 253
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 121 | 110 | 120 | 469
  Male | 34 | 36 | 40 | 25 | 135

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain.
Time Frame: Baseline, Week 16
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Here 'overall number of participants analyzed' signifies participants evaluable for this measure. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 6.06 (1.23) | 5.78 (1.36) | 5.76 (1.32) | 5.87 (1.30)
  Change at Week 16 | -1.91 (1.90) | -2.18 (1.90) | -2.28 (1.99) | -2.42 (2.09)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; LS means were estimated from the corresponding analysis of covariance (ANCOVA) model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.039, ANCOVA; Least Squares (LS) Mean Difference = -0.42, 95% CI 2-sided [-0.81 to -0.02], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; LS means were estimated from the corresponding ANCOVA model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.011, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.91 to -0.12], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.97 to -0.17], Standard Error of Mean 0.20

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 16
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC physical function is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 17 individual questions, each scored on a NRS of 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Here 'overall number of participants analyzed' signifies participants evaluable for this measure. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 157 | 150 | 145
units on a scale
  Baseline | 6.24 (1.45) | 5.86 (1.51) | 5.90 (1.22) | 5.91 (1.36)
  Change at Week 16 | -1.76 (1.78) | -2.11 (1.99) | -2.23 (1.99) | -2.35 (2.07)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.010, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.91 to -0.12], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-1.03 to -0.23], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.10 to -0.30], Standard Error of Mean 0.20

3. Primary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis Score at Week 16
Description: Participants answered: "Considering all the ways your osteoarthritis in your index joint (knee/hip) affects you, how are you doing today?" Participants responded by using a 5-point Likert scale, where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated worst condition.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 3.39 (0.57) | 3.28 (0.46) | 3.43 (0.56) | 3.37 (0.55)
  Change at Week 16 | -0.41 (0.70) | -0.49 (0.74) | -0.61 (0.83) | -0.63 (0.87)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.022, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.32 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.020, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.33 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.40 to -0.09], Standard Error of Mean 0.08

4. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 8, 12 and 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Change at Week 2 | -1.30 (1.43) | -1.22 (1.52) | -1.21 (1.67) | -0.86 (1.57)
  Change at Week 4 | -1.51 (1.55) | -1.76 (1.65) | -2.12 (1.70) | -1.93 (1.71)
  Change at Week 8 | -1.63 (1.54) | -1.88 (1.68) | -2.22 (1.92) | -2.34 (1.92)
  Change at Week 12 | -1.81 (1.59) | -2.23 (1.82) | -2.50 (2.03) | -2.42 (2.00)
  Change at Week 24 | -1.81 (1.91) | -2.11 (2.08) | -2.24 (2.23) | -2.19 (2.16)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; At Week 2: LS means were estimated from the corresponding ANCOVA model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.957, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.32 to 0.34], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.899, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.31 to 0.35], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.022, ANCOVA; LS Mean Difference = 0.39, 95% CI 2-sided [0.06 to 0.72], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; At Week 4: LS means were estimated from the corresponding ANCOVA model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.052, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.70 to 0.00], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.05 to -0.34], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.84 to -0.13], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; At Week 8: LS means were estimated from the corresponding ANCOVA model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.058, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.72 to 0.01], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.05 to -0.32], Standard Error of Mean 0.19
Statistical Analysis 9: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.12 to -0.38], Standard Error of Mean 0.19
Statistical Analysis 10: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; At Week 12: LS means were estimated from the corresponding ANCOVA model. The ANCOVA model included treatment as main effect, baseline value, and index joint as covariates and study site as random effect; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.91 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.80, 95% CI 2-sided [-1.18 to -0.41], Standard Error of Mean 0.20
Statistical Analysis 12: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.05 to -0.28], Standard Error of Mean 0.20

5. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 2, 4, 8, 12, and 24
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Change at Week 2 | -1.31 (1.42) | -1.18 (1.45) | -1.30 (1.57) | -1.06 (1.40)
  Change at Week 4 | -1.46 (1.49) | -1.58 (1.71) | -2.09 (1.84) | -1.81 (1.68)
  Change at Week 8 | -1.59 (1.52) | -1.76 (1.72) | -2.22 (1.88) | -2.13 (1.91)
  Change at Week 12 | -1.75 (1.60) | -2.13 (1.87) | -2.43 (2.01) | -2.28 (1.93)
  Change at Week 24 | -1.70 (1.86) | -1.99 (2.13) | -2.17 (2.19) | -2.08 (2.21)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.754, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.25 to 0.35], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.706, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.36 to 0.25], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.266, ANCOVA; LS Mean Difference = 0.17, 95% CI 2-sided [-0.13 to 0.48], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.195, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.58 to 0.12], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.07 to -0.36], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.019, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.78 to -0.07], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.126, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.64 to 0.08], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.73, 95% CI 2-sided [-1.10 to -0.37], Standard Error of Mean 0.19
Statistical Analysis 9: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.62, 95% CI 2-sided [-0.98 to -0.25], Standard Error of Mean 0.19
Statistical Analysis 10: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.90 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.82, 95% CI 2-sided [-1.21 to -0.44], Standard Error of Mean 0.19
Statistical Analysis 12: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-1.02 to -0.25], Standard Error of Mean 0.20

6. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis Score at Weeks 2, 4, 8, 12, and 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Change at Week 2 | -0.36 (0.79) | -0.37 (0.65) | -0.40 (0.68) | -0.28 (0.71)
  Change at Week 4 | -0.40 (0.74) | -0.45 (0.63) | -0.65 (0.82) | -0.54 (0.75)
  Change at Week 8 | -0.37 (0.72) | -0.44 (0.70) | -0.71 (0.85) | -0.66 (0.79)
  Change at Week 12 | -0.45 (0.80) | -0.52 (0.71) | -0.69 (0.78) | -0.61 (0.76)
  Change at Week 24 | -0.45 (0.77) | -0.46 (0.76) | -0.57 (0.86) | -0.57 (0.91)
Statistical Analysis 1: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.200, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.22 to 0.05], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.754, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.15 to 0.11], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.449, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.08 to 0.18], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.27 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.36 to -0.08], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.026, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.30 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.31 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.48 to -0.19], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.45 to -0.16], Standard Error of Mean 0.08
Statistical Analysis 10: Comparison: Placebo + Diclofenac vs Tanezumab 2.5 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.038, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.30 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 11: Comparison: Placebo + Diclofenac vs Tanezumab 5 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.37 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 12: Comparison: Placebo + Diclofenac vs Tanezumab 10 mg + Diclofenac; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.33 to -0.03], Standard Error of Mean 0.08

7. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response; LOCF
Description: OMERACT-OARSI responder: participant has >=50 percent (%) change and >=2 absolute change from Baseline in either WOMAC pain or physical function subscale scores or at least 2 of the following being true: >=20% change and >=1 absolute change from Baseline in WOMAC pain subscale; >=20% change and >=1 absolute change from Baseline in the WOMAC physical function subscale; >=20% change and >=1 absolute change from Baseline in PGA of osteoarthritis. WOMAC pain and physical function score: 0 to 10 with higher score = worse response. PGA score: 1 = very good and 5 = very poor.
Time Frame: Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
percentage of participants
  Week 2 | 44.7 | 37.2 | 43.3 | 34.5
  Week 4 | 51.3 | 57.1 | 65.3 | 59.3
  Week 8 | 57.2 | 58.3 | 68.0 | 69.7
  Week 12 | 60.5 | 67.3 | 73.3 | 73.1
  Week 16 | 57.9 | 66.7 | 66.7 | 72.4
  Week 24 | 55.3 | 65.4 | 64.7 | 67.6

8. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16 and 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Greater percentage reduction indicates greater improvement. Percentage of participants with cumulative reduction (as percent) (greater than 0%; >= 10, 20, 30, 40, 50, 60, 70, 80 and 90%; = 100 %) in WOMAC pain subscale from Baseline to Weeks 16 and 24 were reported.
Time Frame: Baseline, Week 16 and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Here ' overall number of participants analyzed' signifies participants evaluable for this measure. LOCF method was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
percentage of participants
  Week 16: Greater than 0% reduction | 84.2 | 88.5 | 88.7 | 84.1
  Week 16: >=10% reduction | 73.7 | 82.7 | 76.7 | 77.9
  Week 16: >=20% reduction | 61.8 | 69.9 | 68.7 | 75.2
  Week 16: >=30% reduction | 50.0 | 54.5 | 61.3 | 66.2
  Week 16: >=40% reduction | 38.8 | 48.7 | 50.7 | 60.7
  Week 16: >=50% reduction | 30.9 | 35.9 | 40.0 | 49.0
  Week 16: >=60% reduction | 21.7 | 26.3 | 28.7 | 31.7
  Week 16: >=70% reduction | 13.2 | 17.3 | 20.0 | 19.3
  Week 16: >=80% reduction | 5.9 | 9.0 | 10.7 | 13.8
  Week 16: >=90% reduction | 2.0 | 5.8 | 6.7 | 6.9
  Week 16: 100% reduction | 0.7 | 2.6 | 2.0 | 2.8
  Week 24: Greater than 0% reduction | 81.6 | 82.7 | 82.0 | 84.8
  Week 24: >=10% reduction | 72.4 | 76.9 | 74.7 | 75.2
  Week 24: >=20% reduction | 60.5 | 67.3 | 65.3 | 69.7
  Week 24: >=30% reduction | 48.0 | 58.3 | 59.3 | 59.3
  Week 24: >=40% reduction | 35.5 | 47.4 | 47.3 | 51.0
  Week 24: >=50% reduction | 28.3 | 38.5 | 40.0 | 42.1
  Week 24: >=60% reduction | 20.4 | 26.3 | 34.0 | 31.7
  Week 24: >=70% reduction | 12.5 | 18.6 | 22.7 | 21.4
  Week 24: >=80% reduction | 6.6 | 11.5 | 14.7 | 13.8
  Week 24: >=90% reduction | 3.9 | 8.3 | 8.0 | 8.3
  Week 24: 100% reduction | 0.7 | 3.8 | 3.3 | 2.8

9. Secondary Outcome: Percentage of Participants With At Least 30%, 50%, 70% and 90% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score; LOCF
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Greater percentage reduction indicates greater improvement. Percentage of participants with reduction in WOMAC pain intensity of at least (>=) 30%, 50%, 70% and 90% at Weeks 2, 4, 8, 12, 16, 24 and 32 compared to baseline were classified as responders to WOMAC pain subscale and are reported here.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
percentage of participants
  Week 2: At least 30% reduction | 30.3 | 28.8 | 32.0 | 24.1
  Week 2: At least 50% reduction | 13.8 | 16.0 | 16.7 | 9.0
  Week 2: At least 70% reduction | 4.6 | 6.4 | 7.3 | 2.8
  Week 2: At least 90% reduction | 2.0 | 1.3 | 1.3 | 0.7
  Week 4: At least 30% reduction | 42.1 | 51.9 | 57.3 | 50.3
  Week 4: At least 50% reduction | 17.1 | 26.9 | 34.0 | 30.3
  Week 4: At least 70% reduction | 5.9 | 10.3 | 12.7 | 11.7
  Week 4: At least 90% reduction | 2.0 | 1.9 | 6.0 | 2.1
  Week 8: At least 30% reduction | 43.4 | 51.9 | 57.3 | 63.4
  Week 8: At least 50% reduction | 25.0 | 27.6 | 38.0 | 38.6
  Week 8: At least 70% reduction | 3.9 | 9.6 | 17.3 | 19.3
  Week 8: At least 90% reduction | 2.0 | 5.1 | 4.7 | 6.2
  Week 12: At least 30% reduction | 48.7 | 57.1 | 64.0 | 63.4
  Week 12: At least 50% reduction | 27.0 | 36.5 | 46.7 | 42.8
  Week 12: At least 70% reduction | 7.2 | 16.7 | 24.0 | 24.8
  Week 12: At least 90% reduction | 2.0 | 6.4 | 8.7 | 4.8
  Week 16: At least 30% reduction | 50.0 | 54.5 | 61.3 | 66.2
  Week 16: At least 50% reduction | 30.9 | 35.9 | 40.0 | 49.0
  Week 16: At least 70% reduction | 13.2 | 17.3 | 20.0 | 19.3
  Week 16: At least 90% reduction | 2.0 | 5.8 | 6.7 | 6.9
  Week 24: At least 30% reduction | 48.0 | 58.3 | 59.3 | 59.3
  Week 24: At least 50% reduction | 28.3 | 38.5 | 40.0 | 42.1
  Week 24: At least 70% reduction | 12.5 | 18.6 | 22.7 | 21.4
  Week 24: At least 90% reduction | 3.9 | 8.3 | 8.0 | 8.3

10. Secondary Outcome: Percentage of Participants With Improvement of at Least 2 Points in Patient Global Assessment (PGA) of Osteoarthritis; LOCF
Description: Participants answered: "Considering all the ways your osteoarthritis in your index joint (knee/hip) affects you, how are you doing today?" Participants responded by using a 5-point Likert scale, where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated worst condition. A decrease of at least 2 points on the 5-point scale relative to baseline value indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
percentage of participants
  Week 2 | 5.9 | 5.8 | 4.7 | 5.5
  Week 4 | 6.6 | 3.2 | 14.7 | 12.4
  Week 8 | 5.3 | 6.4 | 18.0 | 14.5
  Week 12 | 6.6 | 6.4 | 14.0 | 12.4
  Week 16 | 4.6 | 5.8 | 14.7 | 16.6
  Week 24 | 5.9 | 5.8 | 12.7 | 12.4

11. Secondary Outcome: Percentage of Participants With Improvement of at Least 2 Points in Patient Global Assessment (PGA) of Osteoarthritis; Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways your osteoarthritis in your index joint (knee/hip) affects you, how are you doing today?" Participants responded by using a 5-point Likert scale, where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated worst condition. A decrease of at least 2 points on the 5-point scale relative to baseline value indicates improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Here 'overall number of participants analyzed' signifies participants evaluable for this measure. BOCF method was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
percentage of participants
  Week 2 | 5.9 | 5.8 | 4.7 | 5.5
  Week 4 | 6.6 | 3.2 | 14.7 | 11.7
  Week 8 | 5.3 | 6.4 | 17.3 | 13.8
  Week 12 | 6.6 | 6.4 | 13.3 | 10.3
  Week 16 | 4.6 | 5.8 | 14.0 | 14.5
  Week 24 | 5.3 | 4.5 | 10.0 | 9.7

12. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee or Hip at Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24
Description: Participants were asked to assess index joint (knee/hip) pain during the past 24 hours on an 0-10 point integer scale ranging from 0 (no pain) to 10 (worst possible pain). Baseline score was calculated as the mean of the scores in the index joint over the 3 days days in the initial pain assessment period and a weekly mean was calculated using the daily pain scores in the index joint within each study week. The change from Baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score, where negative change indicated an improvement.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 142 | 150 | 141 | 134
units on a scale
  Baseline | 6.31 (1.39) | 6.29 (1.30) | 6.38 (1.48) | 6.34 (1.31)
  Change at Week 1 | -0.55 (1.12) | -0.74 (1.10) | -1.22 (1.49) | -0.96 (1.22)
  Change at Week 2 | -0.95 (1.43) | -0.91 (1.40) | -1.28 (1.76) | -1.03 (1.46)
  Change at Week 3 | -1.19 (1.65) | -1.19 (1.57) | -1.40 (1.73) | -1.08 (1.58)
  Change at Week 4 | -1.28 (1.65) | -1.45 (1.70) | -1.77 (1.74) | -1.44 (1.73)
  Change at Week 6 | -1.38 (1.58) | -1.57 (1.75) | -1.88 (1.96) | -1.69 (1.71)
  Change at Week 8 | -1.41 (1.64) | -1.62 (1.75) | -1.84 (2.00) | -1.80 (1.83)
  Change at Week 10 | -1.41 (1.77) | -1.79 (1.88) | -2.09 (2.13) | -2.06 (1.82)
  Change at Week 12 | -1.49 (1.75) | -1.91 (1.82) | -2.06 (2.19) | -2.06 (1.86)
  Change at Week 16 | -1.53 (1.82) | -1.87 (1.90) | -2.07 (2.25) | -2.15 (2.04)
  Change at Week 20 | -1.61 (1.85) | -1.95 (1.94) | -2.19 (2.34) | -2.15 (2.07)
  Change at Week 24 | -1.65 (1.89) | -1.84 (1.96) | -2.07 (2.31) | -2.03 (2.08)

13. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 2, 4, 8, 12, 16, and 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in index knee or hip during past 48 hours. It is calculated as mean of the scores from 2 individual questions scored on NRS of (no stiffness) to 10 (extreme stiffness), with higher scores indicate higher stiffness. Total score range for WOMAC stiffness subscale score is (no stiffness) to 10 (extreme stiffness), where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of knee/hip. Negative change indicated an improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 5.84 (1.78) | 5.61 (1.85) | 5.51 (1.52) | 5.60 (1.78)
  Change at Week 2 | -1.31 (1.75) | -1.29 (1.82) | -1.38 (1.77) | -1.27 (1.91)
  Change at Week 4 | -1.37 (1.83) | -1.71 (2.14) | -2.21 (2.07) | -2.01 (2.16)
  Change at Week 8 | -1.56 (1.89) | -1.86 (2.07) | -2.20 (2.18) | -2.34 (2.22)
  Change at Week 12 | -1.66 (1.94) | -2.36 (2.16) | -2.42 (2.27) | -2.55 (2.22)
  Change at Week 16 | -1.72 (2.11) | -2.27 (2.33) | -2.15 (2.23) | -2.53 (2.26)
  Change at Week 24 | -1.70 (2.17) | -2.06 (2.35) | -2.08 (2.43) | -2.22 (2.34)

14. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, 16, and 24
Description: WOMAC Index: self-administered, disease-specific 24 item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items), and physical function (17 items) in participants with osteoarthritis of the hip and/or knee. WOMAC average score is the mean of the WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, with higher score indicating worse response. Greater reduction in WOMAC average score indicated greater improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 6.05 (1.31) | 5.75 (1.43) | 5.72 (1.19) | 5.80 (1.32)
  Change at Week 2 | -1.31 (1.36) | -1.23 (1.44) | -1.30 (1.52) | -1.06 (1.45)
  Change at Week 4 | -1.45 (1.47) | -1.68 (1.68) | -2.14 (1.74) | -1.92 (1.70)
  Change at Week 8 | -1.59 (1.51) | -1.83 (1.67) | -2.21 (1.86) | -2.27 (1.84)
  Change at Week 12 | -1.74 (1.56) | -2.24 (1.82) | -2.45 (1.97) | -2.42 (1.89)
  Change at Week 16 | -1.80 (1.78) | -2.19 (1.93) | -2.22 (1.93) | -2.43 (2.00)
  Change at Week 24 | -1.74 (1.83) | -2.05 (2.06) | -2.16 (2.16) | -2.17 (2.09)

15. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 2, 4, 8, 12, 16, and 24
Description: Participants answered the question: "How much pain have you had when walking on a flat surface?" Participants responded by using an 11-point scale where 0 = no pain and 10 = extreme pain. Where 0 is the best response and negative change indicated an improvement.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 6.12 (1.67) | 5.91 (1.74) | 5.81 (1.54) | 5.99 (1.71)
  Change at Week 2 | -1.34 (1.71) | -1.23 (1.76) | -1.07 (1.82) | -0.89 (1.86)
  Change at Week 4 | -1.47 (1.74) | -1.75 (2.07) | -2.01 (1.99) | -1.87 (1.96)
  Change at Week 8 | -1.62 (1.78) | -1.81 (1.84) | -2.05 (2.15) | -2.25 (2.31)
  Change at Week 12 | -1.83 (1.92) | -2.15 (1.94) | -2.35 (2.41) | -2.41 (2.36)
  Change at Week 16 | -1.95 (2.12) | -2.14 (1.99) | -2.09 (2.38) | -2.34 (2.52)
  Change at Week 24 | -1.84 (2.13) | -2.08 (2.38) | -2.09 (2.54) | -2.10 (2.62)

16. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Downstairs at Weeks 2, 4, 8, 12, 16, and 24
Description: Participants answered the question: "How much pain have you had when going up or down the stairs?" Participants responded by using an 11-point scale, where 0 = no pain and 10 = extreme pain. Where 0 is the best response and negative change indicated an improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline | 7.24 (1.57) | 7.04 (1.65) | 7.05 (1.63) | 7.06 (1.62)
  Change at Week 2 | -1.38 (1.83) | -1.49 (1.72) | -1.55 (1.94) | -1.21 (1.78)
  Change at Week 4 | -1.58 (1.89) | -2.10 (2.17) | -2.39 (2.13) | -2.10 (2.01)
  Change at Week 8 | -1.78 (1.81) | -2.15 (2.03) | -2.51 (2.40) | -2.64 (2.32)
  Change at Week 12 | -2.03 (1.98) | -2.54 (2.22) | -2.86 (2.51) | -2.77 (2.36)
  Change at Week 16 | -2.00 (2.13) | -2.54 (2.25) | -2.53 (2.40) | -2.79 (2.36)
  Change at Week 24 | -1.95 (2.24) | -2.44 (2.47) | -2.53 (2.51) | -2.56 (2.50)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12 and 24
Description: SF-36v2 was a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and role limitations due to emotional problems, bodily pain, general health, vitality, and mental health. The total score and the score for a section was an average of the individual question scores, which were scaled 0-100. Higher scores reflected better participant status and positive change indicated an improvement.
Time Frame: Baseline, Week 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline: General Health | 46.37 (17.64) | 49.41 (15.67) | 47.00 (15.79) | 49.31 (16.81)
  Baseline: Physical Function | 33.51 (18.98) | 36.22 (18.90) | 34.70 (16.56) | 36.52 (18.46)
  Baseline: Role Physical | 46.67 (21.79) | 47.44 (20.65) | 48.50 (22.21) | 47.46 (22.31)
  Baseline: Bodily Pain | 32.99 (13.77) | 35.66 (12.43) | 33.95 (14.15) | 35.06 (13.47)
  Baseline: Vitality | 49.08 (17.73) | 52.22 (16.82) | 53.00 (17.89) | 51.29 (18.21)
  Baseline: Social Function | 61.02 (23.59) | 67.63 (23.50) | 65.83 (23.65) | 66.55 (23.29)
  Baseline: Role Emotional | 68.15 (26.16) | 68.96 (24.22) | 68.44 (25.86) | 69.77 (24.82)
  Baseline: Mental Health | 62.80 (20.39) | 66.57 (17.12) | 64.63 (18.13) | 65.48 (17.86)
  Change at Week 12: General Health | 4.67 (16.11) | 5.29 (14.70) | 6.55 (13.94) | 4.96 (16.27)
  Change at Week 12: Physical Function | 7.36 (18.33) | 10.96 (20.84) | 12.83 (22.71) | 9.90 (22.60)
  Change at Week 12: Role Physical | 7.61 (22.23) | 8.81 (23.59) | 7.71 (23.45) | 8.49 (25.63)
  Change at Week 12: Bodily Pain | 8.76 (16.79) | 12.51 (20.98) | 15.18 (21.49) | 12.76 (22.62)
  Change at Week 12: Vitality | 3.80 (14.82) | 4.23 (16.17) | 3.79 (18.57) | 5.34 (18.47)
  Change at Week 12: Social Function | 5.02 (22.39) | 6.25 (20.55) | 4.17 (22.37) | 4.22 (22.59)
  Change at Week 12: Role Emotional | 1.92 (24.98) | 2.24 (24.40) | 2.17 (29.05) | -1.26 (27.15)
  Change at Week 12: Mental Health | 3.13 (15.58) | 1.55 (16.05) | 2.20 (16.18) | 1.66 (16.15)
  Change at Week 24: General Health | 2.41 (16.95) | 4.51 (14.94) | 4.94 (15.57) | 3.08 (18.02)
  Change at Week 24: Physical Function | 6.21 (19.01) | 8.78 (22.64) | 10.50 (22.86) | 8.50 (23.87)
  Change at Week 24: Role Physical | 5.17 (22.95) | 8.41 (22.77) | 6.96 (26.61) | 5.91 (27.38)
  Change at Week 24: Bodily Pain | 9.14 (19.41) | 12.54 (21.40) | 13.27 (24.78) | 11.52 (24.58)
  Change at Week 24: Vitality | 1.66 (16.11) | 2.43 (17.72) | 2.58 (20.02) | 2.76 (21.47)
  Change at Week 24: Social Function | 4.36 (22.85) | 4.09 (24.27) | 3.67 (24.04) | 1.38 (28.15)
  Change at Week 24: Role Emotional | -0.55 (25.48) | 0.69 (23.91) | -1.33 (28.95) | -1.95 (27.43)
  Change at Week 24: Mental Health | 1.27 (16.66) | 2.06 (16.93) | 1.63 (16.10) | 0.45 (18.70)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 12 and 24
Description: SF-36v2: standardized survey evaluating 8 aspects of functional health and wellbeing (physical and social functioning, role limitations due to physical and emotional problems, bodily pain, general health, vitality, mental health). Total score for each aspect were scaled 0-100. Higher scores reflect better participant status and positive change indicated an improvement. For obtaining physical and mental component scores, z-score for each scale=(observed score - mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Week 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
z-score
  Baseline: Physical Component Score | -1.84 (0.67) | -1.76 (0.64) | -1.80 (0.61) | -1.76 (0.61)
  Baseline: Mental Component Score | -0.30 (1.16) | -0.11 (1.05) | -0.17 (1.09) | -0.15 (1.12)
  Change at Week 12: Physical Component Score | 0.35 (0.66) | 0.50 (0.76) | 0.56 (0.73) | 0.51 (0.86)
  Change at Week 12: Mental Component Score | 0.08 (0.92) | 0.01 (0.90) | -0.03 (0.96) | -0.06 (1.00)
  Change at Week 24: Physical Component Score | 0.32 (0.76) | 0.45 (0.76) | 0.50 (0.83) | 0.43 (0.91)
  Change at Week 24: Mental Component Score | -0.03 (0.94) | -0.03 (0.98) | -0.10 (0.94) | -0.14 (1.10)

19. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimension (EQ-5D) Index Score at Week 24
Description: EQ-5D was a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme dysfunction) and a single index value characterizing current health status using a visual analog scale with score ranging from 0 (worst) to 100 (best). EQ-5D summary index was obtained with a formula that weights each level of the dimensions. The index-based score was interpreted along a continuum of 0 (death) to 1 (perfect health). Negative change from baseline represented worsening.
Time Frame: Baseline, Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Here 'overall number of participants analyzed' signifies participants evaluable for this measure and 'number analyzed' signifies number of participants evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
units on a scale
  Baseline: Index Score | 0.45 (0.29) | 0.48 (0.25) | 0.47 (0.26) | 0.47 (0.27)
  Change at Week 24: Index Score: number analyzed (Participants) | 96 | 107 | 104 | 95
  Change at Week 24: Index Score | 0.11 (0.35) | 0.15 (0.29) | 0.14 (0.33) | 0.16 (0.31)

20. Secondary Outcome: Number of Participants With Change From Baseline in European Quality of Life - 5 Dimension (EQ-5D) Individual Health State Profile at Week 24
Description: EQ-5D was a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme dysfunction) and a single index value characterizing current health status using a visual analog scale with score ranging from 0 (worst) to 100 (best). Baseline EQ-5D individual health state profile was determined as number of participants "no dysfunction, moderate or some dysfunction and extreme dysfunction" and change from baseline in EQ-5D individual health state profile was determined as number of participants "improved, no change or worsened".
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 156 | 150 | 145
Participants
  Baseline: Mobility-No Dysfunction | 8 | 7 | 14 | 10
  Baseline: Mobility-Moderate Dysfunction | 143 | 148 | 136 | 135
  Baseline: Mobility-Extreme Dysfunction | 1 | 1 | 0 | 0
  Baseline: Self Care-No Dysfunction | 65 | 61 | 53 | 52
  Baseline: Self Care-Moderate Dysfunction | 87 | 92 | 96 | 92
  Baseline: Self Care-Extreme Dysfunction | 0 | 3 | 1 | 1
  Baseline: Usual Activities-No Dysfunction | 25 | 13 | 20 | 18
  Baseline: Usual Activities-Moderate Dysfunction | 116 | 141 | 126 | 123
  Baseline: Usual Activities-Extreme Dysfunction | 11 | 2 | 4 | 4
  Baseline: Pain/Discomfort-No Dysfunction | 0 | 0 | 2 | 1
  Baseline: Pain/Discomfort-Moderate Dysfunction | 114 | 125 | 115 | 111
  Baseline: Pain/Discomfort-Extreme Dysfunction | 38 | 31 | 33 | 33
  Baseline: Anxiety/Depression-No Dysfunction | 74 | 82 | 70 | 73
  Baseline: Anxiety/Depression-Moderate Dysfunction | 72 | 72 | 75 | 66
  Baseline: Anxiety/Depression-Extreme Dysfunction | 6 | 2 | 5 | 6
  Change at Week 24: Mobility-Improved | 21 | 25 | 30 | 25
  Change at Week 24: Mobility-No Change | 127 | 129 | 114 | 120
  Change at Week 24: Mobility-Worsened | 4 | 2 | 6 | 0
  Change at Week 24: Self Care-Improved | 19 | 33 | 32 | 30
  Change at Week 24: Self Care-No Change | 118 | 112 | 110 | 104
  Change at Week 24: Self Care-Worsened | 15 | 11 | 8 | 11
  Change at Week 24: Usual Activities-Improved | 16 | 27 | 31 | 27
  Change at Week 24: Usual Activities-No Change | 125 | 125 | 106 | 111
  Change at Week 24: Usual Activities-Worsened | 11 | 4 | 13 | 7
  Change at Week 24: Pain/Discomfort-Improved | 28 | 29 | 34 | 33
  Change at Week 24: Pain/Discomfort-No Change | 116 | 125 | 109 | 105
  Change at Week 24: Pain/Discomfort-Worsened | 8 | 2 | 7 | 7
  Change at Week 24: Anxiety/Depression-Improved | 27 | 26 | 28 | 19
  Change at Week 24: Anxiety/Depression-No Change | 106 | 111 | 109 | 107
  Change at Week 24: Anxiety/Depression-Worsened | 19 | 19 | 13 | 19

21. Secondary Outcome: Number of Participants Who Discontinued Due to Lack of Efficacy
Description: Number of participants who discontinued due to lack of efficacy were reported.
Time Frame: Baseline up to end of study (Week 32)
Population: The ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 157 | 150 | 145
Participants | 9 | 3 | 7 | 2

22. Secondary Outcome: Time to Discontinuation (TTD) Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16 and 24
Population: as for outcome 21
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 157 | 150 | 145
days
  Week 16 | NA [NA to NA] — Median and 95% confidence interval (CI) limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy.
  Week 24 | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy. | NA [NA to NA] — Median and 95% CI limits cannot be estimated due to the low number of participants who discontinued due to lack of efficacy.

23. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to 112 days after last intravenous dose (up to Week 32)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 157 | 150 | 145
Participants
  AEs | 53 | 71 | 73 | 72
  SAEs | 8 | 12 | 8 | 10

24. Other Pre Specified Outcome: Number of Participants With Intravenous Doses of Study Medication
Description: Number of participants were reported based on the maximum number of intravenous (IV) doses of either tanezumab or placebo received.
Time Frame: Day 1 up to Week 16
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Number analyzed (Participants) | 152 | 157 | 150 | 145
Participants
  Number of IV Doses: 1 | 14 | 9 | 15 | 13
  Number of IV Doses: 2 | 38 | 34 | 26 | 31
  Number of IV Doses: 3 | 100 | 114 | 109 | 101

ADVERSE EVENTS:
Description: Cases of osteonecrosis (ON) reported in this and other studies of this program, conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492.
Arm/Group | Placebo + Diclofenac | Tanezumab 2.5 mg + Diclofenac | Tanezumab 5 mg + Diclofenac | Tanezumab 10 mg + Diclofenac
Serious Adverse Events (participants affected / at risk) | 8/152 | 12/157 | 8/150 | 10/145
Other Adverse Events (participants affected / at risk) | 38/152 | 36/157 | 48/150 | 46/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Diclofenac (N=152) | Tanezumab 2.5 mg + Diclofenac (N=157) | Tanezumab 5 mg + Diclofenac (N=150) | Tanezumab 10 mg + Diclofenac (N=145)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Benign familial pemphigus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Diclofenac (N=152) | Tanezumab 2.5 mg + Diclofenac (N=157) | Tanezumab 5 mg + Diclofenac (N=150) | Tanezumab 10 mg + Diclofenac (N=145)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2 | 3
Toothache (Gastrointestinal disorders) | 9 | 3 | 6 | 1
Oedema peripheral (General disorders) | 2 | 2 | 4 | 7
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 3
Influenza (Infections and infestations) | 1 | 2 | 4 | 2
Nasopharyngitis (Infections and infestations) | 7 | 10 | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7 | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 3
Headache (Nervous system disorders) | 11 | 9 | 7 | 6
Paraesthesia (Nervous system disorders) | 0 | 4 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 3 | 3
Hypertension (Vascular disorders) | 9 | 1 | 3 | 6

LIMITATIONS AND CAVEATS:
Due to United States Food and Drug Administration (FDA) imposed clinical hold, further study drug dosing was stopped prematurely and study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.